CLINICAL TRIAL: NCT02599324
Title: A Phase 1b/2 Study of Ibrutinib Combination Therapy in Selected Advanced Gastrointestinal and Genitourinary Tumors
Brief Title: Study to Evaluate Ibrutinib Combination Therapy in Patients With Selected Gastrointestinal and Genitourinary Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1128-CA; 2015-003656-40 (EudraCT Number)
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Results first posted 2022-10-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-09

CONDITIONS: Metastatic Renal Cell Carcinoma; Advanced Urothelial Carcinoma; Advanced Gastric Adenocarcinoma; Metastatic Colorectal Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — ibrutinib; Everolimus; Paclitaxel; Docetaxel; Cetuximab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1: Renal Cell Carcinoma (RCC) (Experimental): Phase 1b: Participants receive ibrutinib at various dose levels in combination with a fixed dose of everolimus to determine the recommended phase 2 dose (RP2D) of ibrutinib. (The RP2D was determined for each cohort separately.)
  Phase 2: Participants receive ibrutinib at the RP2D determined in phase 1b in combination with everolimus.
  Interventions: Drug: ibrutinib; Drug: everolimus
- Cohort 2: Urothelial Carcinoma (UC) (Experimental): Phase 1b: Participants receive ibrutinib at various dose levels in combination with a fixed dose of paclitaxel to determine the RP2D of ibrutinib. (The RP2D was determined for each cohort separately.)
  Phase 2: Participants receive ibrutinib at the RP2D determined in Phase 1b in combination with paclitaxel.
  Interventions: Drug: ibrutinib; Drug: paclitaxel
- Cohort 3: Gastric Adenocarcinoma (GA or GC) (Experimental): Phase 1b: Participants receive ibrutinib at various dose levels in combination with a fixed dose of docetaxel to determine the RP2D of ibrutinib. (The RP2D was determined for each cohort separately.)
  Phase 2: Participants receive docetaxel at the RP2D determined in Phase 1b in combination with docetaxel.
  Interventions: Drug: ibrutinib; Drug: docetaxel
- Cohort 4: Colorectal Adenocarcinoma (CRC) (Experimental): Phase 1b: Participants receive ibrutinib at various dose levels in combination with a fixed dose of cetuximab to determine RP2D of ibrutinib. (The RP2D was determined for each cohort separately.)
  Phase 2: Participants receive ibrutinib at the RP2D determined in Phase 1b in combination with cetuximab.
  Interventions: Drug: ibrutinib; Drug: cetuximab
- Cohort 5: Urothelial Carcinoma (UC) Ibrutinib (Experimental): Phase 1b: Participants receive ibrutinib at various dose levels to determine the RP2D of ibrutinib.(The RP2D was determined for each cohort separately.)
  Phase 2: Participants receive ibrutinib at the RP2D determined in Phase 1b.
  Interventions: Drug: ibrutinib
- Cohort 6: Urothelial Carcinoma (UC) With Pembrolizumab (Experimental): Phase 1b: Participants receive ibrutinib at various dose levels in combination with a fixed dose of pembrolizumab to determine the RP2D of ibrutinib. (The RP2D was determined for each cohort separately.)
  Phase 2: Participants receive ibrutinib at the RP2D determined in Phase 1b in combination with pembrolizumab.
  Interventions: Drug: ibrutinib; Drug: pembrolizumab

INTERVENTIONS:
Drug: ibrutinib — Ibrutinib administered orally once daily with 8 ounces (approximately 240 mL) of water.
Drug: everolimus — Everolimus 10 mg tablets should be taken orally once daily at the same time every day, either consistently with food or consistently without food. Four (4) x 2.5 mg tablets or two (2) x 5.0 mg tablets may be substituted if 10 mg tablet strength is not available.
  Arms: Cohort 1: Renal Cell Carcinoma (RCC)
Drug: paclitaxel — Paclitaxel should be administered as a 60-minute (±10 minutes) infusion. Paclitaxel should be given at a dose level of 80 mg/m^2, once weekly, in continual 3 weekly cycles.
  Arms: Cohort 2: Urothelial Carcinoma (UC)
Drug: docetaxel — Docetaxel administered as a 60 minute infusion (±10 minutes) at a dose level of 60 - 75 mg/m^2 (according to local institutional standard of care), given continually in 21-day cycles.
  Arms: Cohort 3: Gastric Adenocarcinoma (GA or GC)
Drug: cetuximab — Cetuximab 400 mg/m^2 administered as a 120-minute IV infusion. The recommended subsequent weekly dose (all other infusions) is 250 mg/m^2 infused over 60 minutes.
  Arms: Cohort 4: Colorectal Adenocarcinoma (CRC)
Drug: pembrolizumab — Pembrolizumab 200 mg intravenous (IV) every 3 weeks.
  Arms: Cohort 6: Urothelial Carcinoma (UC) With Pembrolizumab

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of single agent ibrutinib or the combination treatments of ibrutinib with everolimus, paclitaxel, docetaxel, pembrolizumab or cetuximab in selected advance gastrointestinal and genitourinary tumors.

ELIGIBILITY:
Inclusion Criteria:

RCC (clear cell), urothelial carcinoma (UC) (transitional cell), gastric or gastro-esophageal junctional (GEJ) adenocarcinoma, or K-RAS or N-RAS wild-type EGFR expressing CRC For cohort 1 RCC: minimum of 1 and maximum of 4 prior regimens, one or more of which must have included a VEGF-TKI For UC cohort 2: minimum of 1 and maximum of 2 prior regimens, one of which must have included a platinum-based regimen For UC cohort 5: Minimum of 1 and maximum of 2 prior regimens, one of which must have included a checkpoint inhibitor.

For UC cohort 6:

Locally advanced or mUC who are not eligible for cisplatin chemo with a PDL-1 score (CPS) of ≥ 10 without prior treatment.

Locally advanced or mUC who have progressed on platinum chemo or within 12 months of neo- or adjuvant therapy with a platinum chemotherapy. A minimum of 1 and maximum of 2 prior therapies.

For cohort 3 gastric or GEJ adenocarcinoma: minimum of 1 and maximum of 3 prior regimens one of which must have included a fluoropyrimidine regimen For cohort 4 CRC: minimum of 2 and maximum of 4 prior regimens, which must have included both an irinotecan and an oxaliplatin based regimen unless unable to tolerate irinotecan chemotherapy

Laboratory:

Adequate hematologic function:

Absolute neutrophil count ≥1500 cells/mm3 (1.5 x 109/L) Platelet count >80,000 cells/mm3 (80 x 109/L) for cohort 1 (RCC) Platelet counts >100,000 cells/mm3 (100 x 109/L) for all UC cohorts Hemoglobin ≥8.0 g/dL. for cohort 1 (RCC),all UC cohorts, and cohort 3 (GC) Hemoglobin ≥9.0 g/dL for cohort 4 (CRC)

Adequate hepatic and renal function defined as:

Serum aspartate transaminase (AST) and/or alanine transaminase (ALT) ≤5.0 x upper limit of normal (ULN) if liver metastases, or ≤3 x ULN without liver metastases Alkaline phosphatase <3.0 x ULN or ≤5.0 x ULN if liver or bone metastases present Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin, such as hemolysis) with the exception of subjects in the GC cohort where docetaxel is administered, these subjects must have bilirubin within normal limits (WNL) Estimated Creatinine Clearance ≥30 mL/min (Cockcroft-Gault)

Exclusion Criteria

Prior treatment with:

Everolimus or temsirolimus (RCC cohort 1) Any taxane (UC cohort of ibrutinib + paclitaxel) (cohort 2) Checkpoint inhibitors (UC cohort 6) Any taxane (GC cohort 3) Cetuximab or panitumumab (CRC cohort 4)

For all Cohorts:

Concomitant use of warfarin or other Vitamin K antagonists History of stroke or intracranial hemorrhage within 6 months prior to enrollment Major surgery within 4 weeks of first dose of study drug Requires treatment with strong CYP3A inhibitors known bleeding disorders or hemophilia

UC cohort 6 only:

Subjects who have an active, known or suspected autoimmune disease. Evidence of clinically significant interstitial lung disease or active, noninfectious pneumonitis.

Non-steroid immunosuppressive medications within 14 days before the first dose of ibrutinib and pembrolizumab.

Subjects in whom prior anti PD-1 / anti-PD-L1 therapy was intolerable and required discontinuation of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pharmacyclics LLC, Study Director — Pharmacyclics LLC.
Locations (65):
- United States (44):
  - Clearview Cancer Institute /ID# 1128-0965, Huntsville, Alabama
  - Banner MD Anderson Cancer Center /ID# 1128-0802, Gilbert, Arizona
  - University of Arizona Cancer Center - Tucson /ID# 1128-1546, Tucson, Arizona
  - Alta Bates Comprehensive Cancer Center /ID# 1128-0135, Berkeley, California
  - St Marys Medical Center /ID# 1128-0969, Daly City, California
  - Duplicate_University of California San Diego/ Moores Cancer Center /ID# 1128-0241, La Jolla, California
  - VA Long Beach Healthcare System /ID# 1128-0480, Long Beach, California
  - USC Norris Cancer Center /ID# 1128-0209, Los Angeles, California
  - UC Irvine Medical Center - Chao Family Comprehensive Cancer Center /ID# 1128-0008, Orange, California
  - Salinas Valley Memorial Hosp /ID# 1128-0482, Salinas, California
  - Premiere Oncology, A Medical Corporation /ID# 1128-1085, Santa Monica, California
  - St. Joseph Health /ID# 1128-1462, Santa Rosa, California
  - Gregory Smith, MD (Private Practice) /ID# 1128-0419, St. Helena, California
  - Whittingham Cancer Center at Norwalk Hospital /ID# 1128-0411, Norwalk, Connecticut
  - Georgetown University Hospital /ID# 1128-0824, Washington D.C., District of Columbia
  - Duplicate_Cancer Specialist of North Florida (CSNF) ( R ) /ID# 1128-1093, Jacksonville, Florida
  - IACT Health-Columbus /ID# 1128-1389, Columbus, Georgia
  - Northshore Kellogg Cancer Center /ID# 1128-0484, Evanston, Illinois
  - Franciscan Health Indianapolis /ID# 1128-1125, Indianapolis, Indiana
  - Horizon Oncology Research Center /ID# 1128-0337, Lafayette, Indiana
  - University of Iowa Hospitals and Clinics /ID# 1128-0766, Iowa City, Iowa
  - The University of Kansas Cancer Center /ID# 1128-0706, Fairway, Kansas
  - East Jefferson General Hospital /ID# 1128-1084, Metairie, Louisiana
  - Duplicate_Tufts Medical Center /ID# 1128-0016, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer In /ID# 1128-0130, Detroit, Michigan
  - Henry Ford Hospital /ID# 1128-0195, Detroit, Michigan
  - Central Care Cancer Center /ID# 1128-1596, Bolivar, Missouri
  - Capital Region Medical Center /ID# 1128-1412, Jefferson City, Missouri
  - Nebraska Methodist Hospital /ID# 1128-0229, Omaha, Nebraska
  - New Jersey Center for Cancer Research /ID# 1128-0493, Brick, New Jersey
  - Duplicate_New Mexico Cancer Care Alliance /ID# 1128-0938, Albuquerque, New Mexico
  - San Juan Oncology Associates /ID# 1128-1020, Farmington, New Mexico
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 1128-0091, New York, New York
  - Wake Forest Univ HS /ID# 1128-0975, Winston-Salem, North Carolina
  - Oregon Health & Science University /ID# 1128-0251, Portland, Oregon
  - Penn State Hershey Medical Ctr /ID# 1128-0220, Hershey, Pennsylvania
  - Abramson Cancer Center of the Univ. of Pennsylvania /ID# 1128-0402, Philadelphia, Pennsylvania
  - Vanderbilt Infectious Disease Clinic /ID# 1128-0024, Nashville, Tennessee
  - The University of Texas Medical Branch (UTMB) - Cancer Center - Galves /ID# 1128-0974, Galveston, Texas
  - Duplicate_Scott & White Mem Hosp & Clin /ID# 1128-0046, Temple, Texas
  - Duplicate_Virginia Cancer Specialists - Fairfax Office /ID# 1128-0972, Fairfax, Virginia
  - Virginia Mason Medical Center /ID# 1128-0005, Seattle, Washington
  - University of Washington /ID# 1128-1382, Seattle, Washington
  - Confluence Health /ID# 1128-0894, Wenatchee, Washington
- South Korea (8):
  - Seoul National University Bundang Hospital /ID# 1128-0982, Seongnam, Gyeonggido
  - Yonsei University Health System Severance Hospital /ID# 1128-0927, Seoul, Seoul Teugbyeolsi
  - Chonnam National University Hwasun Hospital /ID# 1128-0916, Jeonnam
  - Seoul National University Hospital /ID# 1128-0926, Seoul
  - Asan Medical Center /ID# 1128-0963, Seoul
  - Samsung Medical Center /ID# 1128-0925, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital /ID# 1128-0928, Seoul
  - Korea University Guro Hospital /ID# 1128-0924, Seoul
- Spain (8):
  - Instituto Catalan de Oncologia (ICO) Badalona /ID# 1128-0984, Badalona, Barcelona
  - Hospital Unversitario Marques de Valdecilla /ID# 1128-0973, Santander, Cantabria
  - Hospital Universitario Vall d'Hebron /ID# 1128-0534, Barcelona
  - Hospital Clinic de Barcelona /ID# 1128-0533, Barcelona
  - Hospital Universitario Ramon y Cajal /ID# 1128-0874, Madrid
  - Hospital Universitario 12 de Octubre /ID# 1128-0864, Madrid
  - Hospital Universitario La Paz /ID# 1128-0921, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 1128-0863, Seville
- United Kingdom (5):
  - Sarah Cannon Research Institute /ID# 1128-1079, London, England
  - Duplicate_Beatson west of scotland cancer center /ID# 1128-0652, Glasgow, Scotland
  - The Royal Marsden NHS Foundation Trust /ID# 1128-0543, London
  - The Christie Hospital /ID# 1128-0030, Manchester
  - Duplicate_Oxford University Hospitals NHS Trust /ID# 1128-0814, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Requests for access to individual participant data from clinical studies conducted by Pharmacyclics LLC, an AbbVie Company, can be submitted through Yale Open Data Access (YODA) Project site at the following link.
Supporting Information: Study Protocol, SAP, CSR
URL: http://yoda.yale.edu

REFERENCES:
- [Derived] Oh DY, Maqueda MA, Quinn DI, O'Dwyer PJ, Chau I, Kim SY, Duran I, Castellano D, Berlin J, Mellado B, Williamson SK, Lee KW, Marti F, Mathew P, Saif MW, Wang D, Chong E, Hilger-Rolfe J, Dean JP, Arkenau HT. Ibrutinib combination therapy for advanced gastrointestinal and genitourinary tumours: results from a phase 1b/2 study. BMC Cancer. 2023 Nov 3;23(1):1056. doi: 10.1186/s12885-023-11539-1. PMID 37919668

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Phase 1b, participants were enrolled into 6 separate cohorts according to clinical indication: renal cell carcinoma (RCC; Cohort 1), urothelial carcinoma (UC; Cohort 2), gastric adenocarcinoma (GA; Cohort 3), colorectal adenocarcinoma (CRC; Cohort 4), urothelial carcinoma (UC; Cohorts 5 and 6). A dose level review committee (DLRC) evaluated the safety data at the completion of Phase 1b in each cohort to determine the recommended Phase 2 dose (RP2D), with the exception of Cohort 5.
Pre-assignment Details: For Cohorts 1 to 4 and 6, participants enrolled into 5 distinct disease specific cohorts to receive ibrutinib at the RP2D determined in Phase 1b for that cohort in combination with the relative cancer agent. Treatment was to follow the same dosing schedule used in Phase 1b, and all cohorts were to continue on ibrutinib RP2D and respective anticancer agents until disease progression or unacceptable toxicity. For Cohort 5, single agent ibrutinib was given at the RP2D PO daily in 21-day cycles.
Groups:
- Cohort 1 (RCC): Ibrutinib 560 mg + Everolimus: Phase 1b: Participants with RCC received ibrutinib 560 mg once daily (QD) in combination with everolimus 10 mg QD.
- Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus: Phase 1b: Participants with RCC received ibrutinib 840 mg QD in combination with everolimus 10 mg QD.
  Phase 2 (RP2D): Participants with RCC received ibrutinib 840 mg QD in combination with everolimus 10 mg QD.
- Cohort 2 (UC): Ibrutinib 560 mg + Paclitaxel: Phase 1b: Participants with UC received ibrutinib 560 mg QD in combination with paclitaxel 80 mg/m^2, once weekly, in continual 3 weekly cycles.
- Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel: Phase 1b: Participants with UC received ibrutinib 840 mg QD in combination with paclitaxel 80 mg/m^2, once weekly, in continual 3 weekly cycles.
  Phase 2 (RP2D): Participants with UC received ibrutinib 840 mg QD in combination with paclitaxel 80 mg/m^2, once weekly, in continual 3 weekly cycles.
- Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel: Phase 1b: Participants with GA received ibrutinib 560 mg QD in combination with docetaxel administered as a 60 minute infusion (±10 minutes) at a dose level of 60 - 75 mg/m^2, given continually in 21 day cycles.
  Phase 2 (RP2D): Participants with GA received ibrutinib 560 mg QD in combination with docetaxel administered as a 60 minute infusion (±10 minutes) at a dose level of 60 - 75 mg/m^2, given continually in 21 day cycles.
- Cohort 4 (CRC): Ibrutinib 560 mg + Cetuximab: Phase 1b: Participants with CRC received ibrutinib 560 mg QD in combination with cetuximab 400 mg/m^2 administered as a 120-minute IV infusion. Subsequent weekly dose (all other infusions) was 250 mg/m^2 infused over 60 minutes.
- Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab: Phase 1b: Participants with CRC received ibrutinib 840 mg QD in combination with cetuximab 400 mg/m^2 administered as a 120-minute IV infusion. Subsequent weekly dose (all other infusions) was 250 mg/m^2 infused over 60 minutes.
  Phase 2 (RP2D): Participants with CRC received ibrutinib 840 mg QD in combination with cetuximab 400 mg/m^2 administered as a 120-minute IV infusion. Subsequent weekly dose (all other infusions) was 250 mg/m^2 infused over 60 minutes.
- Cohort 5 (UC): Ibrutinib 840 mg: Phase 1b: Participants with UC received monotherapy with ibrutinib 840 mg QD.
  Phase 2 (RP2D): Participants with UC received monotherapy with ibrutinib 840 mg QD.
- Cohort 6 (UC): Ibrutinib 560 mg + Pembrolizumab: Phase 1b: Participants with UC received ibrutinib 560 mg QD in combination with pembrolizumab 200 mg IV every 3 weeks.
  Phase 2 (RP2D): Participants with UC received ibrutinib 560 mg QD in combination with pembrolizumab 200 mg IV every 3 weeks.
Period: Phase 1b
Arm/Group | Cohort 1 (RCC): Ibrutinib 560 mg + Everolimus | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 560 mg + Paclitaxel | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 560 mg + Cetuximab | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab | Cohort 5 (UC): Ibrutinib 840 mg | Cohort 6 (UC): Ibrutinib 560 mg + Pembrolizumab
Started | 3 | 7 | 4 | 10 | 21 | 8 | 12 | 10 | 17
Completed | 3 | 7 | 4 | 10 | 21 | 8 | 12 | 10 | 17
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2 (RP2D)
Arm/Group | Cohort 1 (RCC): Ibrutinib 560 mg + Everolimus | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 560 mg + Paclitaxel | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 560 mg + Cetuximab | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab | Cohort 5 (UC): Ibrutinib 840 mg | Cohort 6 (UC): Ibrutinib 560 mg + Pembrolizumab
Started (Entered Phase 2 and received at least 1 dose of study medication.) | 0 | 38 | 0 | 55 | 31 | 0 | 44 | 33 | 13
Continued From Phase 1b | 0 | 6 | 0 | 6 | 6 | 0 | 6 | 8 | 12
Enrolled in Phase 2 | 0 | 32 | 0 | 49 | 25 | 0 | 39 | 25 | 1
Enrolled and Treated in Phase 2 | 0 | 32 | 0 | 49 | 25 | 0 | 38 | 25 | 1
Completed (Off Study) | 0 | 38 | 0 | 55 | 31 | 0 | 44 | 33 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated population: all unique participants enrolled and treated in Phase 1b and Phase 2.
Groups:
- Cohort 1 (RCC): Ibrutinib 560 mg + Everolimus: Participants with RCC received ibrutinib 560 mg QD in combination with everolimus 10 mg QD.
- Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus: Participants with RCC received ibrutinib 840 mg QD in combination with everolimus 10 mg QD.
- Cohort 2 (UC): Ibrutinib 560 mg + Paclitaxel: Participants with UC received ibrutinib 560 mg QD in combination with paclitaxel 80 mg/m^2, once weekly, in continual 3 weekly cycles.
- Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel: Participants with UC received ibrutinib 840 mg QD in combination with paclitaxel 80 mg/m^2, once weekly, in continual 3 weekly cycles.
- Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel: Participants with GA received ibrutinib 560 mg QD in combination with docetaxel administered as a 60 minute infusion (±10 minutes) at a dose level of 60 - 75 mg/m^2, given continually in 21 day cycles.
- Cohort 4 (CRC): Ibrutinib 560 mg + Cetuximab: Participants with CRC received ibrutinib 560 mg QD in combination with cetuximab 400 mg/m^2 administered as a 120-minute IV infusion. Subsequent weekly dose (all other infusions) was 250 mg/m^2 infused over 60 minutes.
- Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab: Participants with CRC received ibrutinib 840 mg QD in combination with cetuximab 400 mg/m^2 administered as a 120-minute IV infusion. Subsequent weekly dose (all other infusions) was 250 mg/m^2 infused over 60 minutes.
- Cohort 5 (UC): Ibrutinib 840 mg: Participants with UC received monotherapy with ibrutinib 840 mg QD.
- Cohort 6 (UC): Ibrutinib 560 mg + Pembrolizumab: Participants with UC received ibrutinib 560 mg QD in combination with pembrolizumab 200 mg IV every 3 weeks.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (RCC): Ibrutinib 560 mg + Everolimus | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 560 mg + Paclitaxel | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 560 mg + Cetuximab | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab | Cohort 5 (UC): Ibrutinib 840 mg | Cohort 6 (UC): Ibrutinib 560 mg + Pembrolizumab | Total
Number analyzed (Participants) | 3 | 39 | 4 | 59 | 46 | 8 | 50 | 35 | 18 | 262
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 1 | 23 | 3 | 21 | 33 | 6 | 25 | 11 | 6 | 129
  65 - 84 years | 2 | 16 | 1 | 35 | 13 | 2 | 25 | 22 | 12 | 128
  ≥ 85 years | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 0 | 8 | 12 | 7 | 21 | 9 | 5 | 71
  Male | 2 | 31 | 4 | 51 | 34 | 1 | 29 | 26 | 13 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 4 | 7 | 3 | 0 | 1 | 1 | 18
  Not Hispanic or Latino | 3 | 39 | 2 | 55 | 39 | 4 | 50 | 34 | 17 | 243
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 7 | 0 | 12 | 12 | 2 | 31 | 5 | 0 | 69
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 4
  White | 3 | 32 | 4 | 47 | 32 | 5 | 18 | 30 | 16 | 187
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose-Limiting Toxicities (DLTs) in Cohorts 1 to 6
Description: A DLT was defined as any Grade 3 (severe) or higher non-hematologic or Grade 4 (life-threatening) hematologic adverse event (AE) occurring during the DLT observation period that was considered to be at least possibly related to the study treatment (ibrutinib or drug combination).
Time Frame: 21 days after the initiation of therapy at the start of Cycle 1
Population: DLT Evaluable Population: participants from Phase 1b who completed at least 21 days of treatment with ibrutinib in combination with the relevant anticancer agent after the initiation of study treatment at the start of Cycle 1, or those who discontinued from study treatment due to a DLT event prior to completion of DLT observation period. For UC Cohorts 5 and 6, a DLT-evaluable participant had ≥ 90% compliance with ibrutinib during Cycle 1 (the first 21 days).
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 (RCC): Ibrutinib 560 mg + Everolimus: Participants with RCC received ibrutinib 560 mg QD in combination with everolimus 10 mg QD in Phase 1b.
- Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus: Participants with RCC received ibrutinib 840 mg QD in combination with everolimus 10 mg QD in Phase 1b.
- Cohort 2 (UC): Ibrutinib 560 mg + Paclitaxel: Participants with UC received ibrutinib 560 mg QD in combination with paclitaxel 80 mg/m^2, once weekly, in continual 3 weekly cycles in Phase 1b.
- Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel: Participants with UC received ibrutinib 840 mg QD in combination with paclitaxel 80 mg/m^2, once weekly, in continual 3 weekly cycles in Phase 1b.
- Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel: Participants with GA received ibrutinib 560 mg QD in combination with docetaxel administered as a 60 minute infusion (±10 minutes) at a dose level of 60 - 75 mg/m^2, given continually in 21 day cycles Phase 1b.
- Cohort 4 (CRC): Ibrutinib 560 mg + Cetuximab: Participants with CRC received ibrutinib 560 mg QD in combination with cetuximab 400 mg/m^2 administered as a 120-minute IV infusion. Subsequent weekly dose (all other infusions) was 250 mg/m^2 infused over 60 minutes Phase 1b.
- Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab: Participants with CRC received ibrutinib 840 mg QD in combination with cetuximab 400 mg/m^2 administered as a 120-minute IV infusion. Subsequent weekly dose (all other infusions) was 250 mg/m^2 infused over 60 minutes in Phase 1b.
- Cohort 5 (UC): Ibrutinib 840 mg: Participants with UC received monotherapy with ibrutinib 840 mg QD in Phase 1b.
- Cohort 6 (UC): Ibrutinib 560 mg + Pembrolizumab: Participants with UC received ibrutinib 560 mg QD in combination with pembrolizumab 200 mg IV every 3 weeks in Phase 1b.
Arm/Group | Cohort 1 (RCC): Ibrutinib 560 mg + Everolimus | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 560 mg + Paclitaxel | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 560 mg + Cetuximab | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab | Cohort 5 (UC): Ibrutinib 840 mg | Cohort 6 (UC): Ibrutinib 560 mg + Pembrolizumab
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 7 | 3 | 6 | 7 | 10
Participants | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 1b/2 RP2D: Progression-Free Survival (PFS) as Assessed by Investigator in Cohorts 1 and 2
Description: PFS is defined as the time from the date of first dose of study treatment to the date of first documentation of progressive disease (PD) or date of death from any cause, whichever occurs first, regardless of the use of subsequent anti-cancer treatment. PD was defined in accordance with Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study), and an absolute increase of ≥ 5 mm, or unequivocal progression of existing non-target lesions or the appearance of new lesions.
Time Frame: Maximum time on study for Cohort 1 (Phase 1b/2 RP2D) was 37.4 months; for Cohort 2 (Phase 1b/2 RP2D) was 44.7 months.
Population: Efficacy Evaluable Population: Participants who received at least one dose of ibrutinib (at RP2D) in combination with at least one dose of the relevant companion drug and had at least one adequate post-baseline overall disease assessment per RECIST 1.1 guidelines or died prior to the first adequate post-baseline overall disease assessment. Per protocol, participants in Phase 1b receiving the Phase 2 RP2D and participants in Phase 2 RP2D were analyzed together.
Measure: Median (90% Confidence Interval); unit: months
Groups:
- Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus: Participants with RCC received ibrutinib 840 mg QD in combination with everolimus 10 mg QD in Phase 1b/2 RP2D.
- Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel: Participants with UC received ibrutinib 840 mg QD in combination with paclitaxel 80 mg/m^2, once weekly, in continual 3 weekly cycles in Phase 1b/2 RP2D.
Arm/Group | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel
Number analyzed (Participants) | 36 | 57
months | 5.6 [3.9 to 7.5] | 4.1 [2.7 to 4.4]

3. Primary Outcome: Phase 1b/2 RP2D: Overall Response Rate (ORR) as Assessed by Investigator in Cohorts 3 to 6
Description: ORR is defined as the percentage of participants who have a best response of partial response (PR) or complete response (CR) to therapy in accordance with RECIST 1.1 criteria. CR: The disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Normalization of tumor marker level, if relevant. All lymph nodes must be non-pathological in size (< 10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Maximum time on study (Phase 1b/2 RP2D) for Cohort 3 was 41.9 months; for Cohort 4 was 23.5 months; for Cohort 5 was 17.3 months; for Cohort 6 was 20.1 months.
Population: Efficacy Evaluable Population (Phase 1b/2 RP2D): participants who received ≥ 1 dose of ibrutinib (at RP2D) in combination with ≥ 1 dose of the relevant companion drug or ibrutinib (at RP2D) for the single-agent therapy and: 1) Had measurable disease per RECIST 1.1 guidelines at baseline. 2) Had ≥ 1 adequate post-baseline overall disease assessment per RECIST 1.1 guidelines. Per protocol, participants in Phase 1b receiving the Phase 2 RP2D and participants in Phase 2 RP2D were analyzed together.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel: Participants with GA received ibrutinib 560 mg QD in combination with docetaxel administered as a 60 minute infusion (±10 minutes) at a dose level of 60 - 75 mg/m^2, given continually in 21 day cycles in Phase 1b/2 RP2D.
- Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab: Participants with CRC received ibrutinib 840 mg QD in combination with cetuximab 400 mg/m^2 administered as a 120-minute IV infusion. Subsequent weekly dose (all other infusions) was 250 mg/m^2 infused over 60 minutes in Phase 1b/2 RP2D.
- Cohort 5 (UC): Ibrutinib 840 mg: Participants with UC received monotherapy with ibrutinib 840 mg QD in Phase 1b/2 RP2D.
- Cohort 6 (UC): Ibrutinib 560 mg + Pembrolizumab: Participants with UC received ibrutinib 560 mg QD in combination with pembrolizumab 200 mg IV every 3 weeks in Phase 1b/2 RP2D.
Arm/Group | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab | Cohort 5 (UC): Ibrutinib 840 mg | Cohort 6 (UC): Ibrutinib 560 mg + Pembrolizumab
Number analyzed (Participants) | 39 | 47 | 29 | 14
percentage of participants | 17.9 [8.7 to 31.1] | 14.9 [7.2 to 26.2] | 6.9 [1.2 to 20.2] | 35.7 [15.3 to 61.0]

4. Secondary Outcome: Phase 1b: ORR in Cohorts 1 to 6
Description: as for outcome 3
Time Frame: Maximum time on study (Phase 1b only) for Cohort 1 was 37.4 months; for Cohort 2 was 44.7 months; for Cohort 3 was 41.9 months; for Cohort 4 was 34.2 months; for Cohort 5 was 17.3 months; for Cohort 6 was 20.1 months.
Population: Efficacy Evaluable Population (Phase 1b): participants who received at least one dose of ibrutinib (at RP2D) in combination with at least one dose of the relevant companion drug or ibrutinib (at RP2D) for the single-agent therapy and: 1) Had measurable disease per RECIST 1.1 guidelines at baseline. 2) Had at least one adequate post-baseline overall disease assessment per RECIST 1.1 guidelines.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (RCC): Ibrutinib 560 mg + Everolimus | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 560 mg + Paclitaxel | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 560 mg + Cetuximab | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab | Cohort 5 (UC): Ibrutinib 840 mg | Cohort 6 (UC): Ibrutinib 560 mg + Pembrolizumab
Number analyzed (Participants) | 3 | 7 | 4 | 10 | 18 | 8 | 10 | 8 | 13
percentage of participants | 0 [0.0 to 63.2] | 0 [0.0 to 34.8] | 50.0 [9.8 to 90.2] | 20.0 [3.7 to 50.7] | 11.1 [2.0 to 31.0] | 12.5 [0.6 to 47.1] | 0 [0.0 to 25.9] | 12.5 [0.6 to 47.1] | 38.5 [16.6 to 64.5]

5. Secondary Outcome: Phase 1b: Disease Control Rate (DCR) in Cohorts 1 to 6
Description: DCR is is defined as the percentage of participants who have a best response of PR, CR, or stable disease (SD) to therapy in accordance with RECIST 1.1 criteria. CR: The disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Normalization of tumor marker level, if relevant. All lymph nodes must be non-pathological in size (< 10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SOD since the treatment started (baseline or after). For SD, tthere was no need for confirmation by a subsequent imaging assessment.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (RCC): Ibrutinib 560 mg + Everolimus | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 560 mg + Paclitaxel | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 560 mg + Cetuximab | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab | Cohort 5 (UC): Ibrutinib 840 mg | Cohort 6 (UC): Ibrutinib 560 mg + Pembrolizumab
Number analyzed (Participants) | 3 | 7 | 4 | 10 | 18 | 8 | 10 | 8 | 13
percentage of participants | 66.7 [13.5 to 98.3] | 71.4 [34.1 to 94.7] | 75.0 [24.9 to 98.7] | 50.0 [22.2 to 77.8] | 77.8 [56.1 to 92.0] | 75.0 [40.0 to 95.4] | 80.0 [49.3 to 96.3] | 37.5 [11.1 to 71.1] | 76.9 [50.5 to 93.4]

6. Secondary Outcome: Phase 1b/2 RP2D: DCR in Cohorts 1 to 6
Description: DCR is is defined as the percentage of participants who have a best response of PR, CR, or SD to therapy in accordance with RECIST 1.1 criteria. CR: The disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Normalization of tumor marker level, if relevant. All lymph nodes must be non-pathological in size (< 10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SOD since the treatment started (baseline or after). For SD, tthere was no need for confirmation by a subsequent imaging assessment.
Time Frame: Maximum time on study (Phase 1b/2 RP2D) for Cohort 1 was 37.4 months; for Cohort 2 was 44.7 months; for Cohort 3 was 41.9 months; for Cohort 4 was 23.5 months; for Cohort 5 was 17.3 months; for Cohort 6 was 20.1 months. (Reverse Kaplan-Meier estimates)
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab | Cohort 5 (UC): Ibrutinib 840 mg | Cohort 6 (UC): Ibrutinib 560 mg + Pembrolizumab
Number analyzed (Participants) | 36 | 57 | 39 | 47 | 29 | 14
percentage of participants | 80.6 [66.6 to 90.5] | 66.7 [55.0 to 77.0] | 74.4 [60.4 to 85.4] | 83.0 [71.4 to 91.2] | 48.3 [32.0 to 64.8] | 71.4 [46.0 to 89.6]

7. Secondary Outcome: Phase 1b/2 RP2D: PFS in Cohorts 3 to 6
Description: PFS is defined as the time from the date of first dose of study treatment to the date of first documentation of PD or date of death from any cause, whichever occurs first, regardless of the use of subsequent anti-cancer treatment. PD was defined in accordance with RECIST 1.1 criteria.
Time Frame: Maximum time on study (Phase 1b/2 RP2D) for Cohort 3 was 41.9 months; for Cohort 4 was 23.5 months; for Cohort 5 was 17.3 months; for Cohort 6 was 20.1 months. (Reverse Kaplan-Meier estimates)
Population: as for outcome 3
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab | Cohort 5 (UC): Ibrutinib 840 mg | Cohort 6 (UC): Ibrutinib 560 mg + Pembrolizumab
Number analyzed (Participants) | 39 | 47 | 29 | 14
months | 4.0 [2.7 to 4.2] | 5.4 [4.1 to 5.8] | 1.6 [1.4 to 2.5] | 2.9 [1.7 to NA] — Not estimable because of the small number of events.

8. Secondary Outcome: Phase 1b/2 RP2D: ORR in Cohorts 1 and 2
Description: ORR is defined as the percentage of participants who have a best response to therapy of PR or CR in accordance with RECIST 1.1 criteria. CR: The disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Normalization of tumor marker level, if relevant. All lymph nodes must be non-pathological in size (< 10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Maximum time on study for Cohort 1 (Phase 1b/2 RP2D) was 37.4 months; for Cohort 2 (Phase 1b/2 RP2D) was 44.7 months. (Reverse Kaplan-Meier estimates)
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel
Number analyzed (Participants) | 36 | 57
percentage of participants | 2.8 [0.1 to 12.5] | 26.3 [17.0 to 37.6]

9. Secondary Outcome: Phase 1b/2 RP2D: Overall Survival (OS) in Cohorts 1 to 6
Description: OS is defined as the time from the date of first dose of study treatment to the date of death from any cause. Subjects who were not known to have died at the data extraction will be censored at date last known alive.
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab | Cohort 5 (UC): Ibrutinib 840 mg | Cohort 6 (UC): Ibrutinib 560 mg + Pembrolizumab
Number analyzed (Participants) | 36 | 57 | 39 | 47 | 29 | 14
months | 21.0 [13.1 to 25.3] | 8.2 [6.2 to 10.3] | 7.3 [5.5 to 9.6] | 15.0 [10.5 to 17.2] | 8.2 [4.4 to NA] — Not estimable because of the small number of events. | 15.7 [7.7 to NA] — Not estimable because of the small number of events.

10. Secondary Outcome: Phase 1b/2 RP2D: Duration of Response (DOR) in Cohorts 1 to 6
Description: DOR is defined for confirmed responders (PR or better) as time from the date of initial response (PR or better) to the date of first documentation of PD (according to RECIST 1.1) or death, whichever occurs first, regardless of use of subsequent anti-cancer treatment. Confirmed responders without documentation of PD or death or with unknown status at the data extraction were censored at the last adequate post-baseline disease assessment showing no evidence of PD. PD was defined as at least a 20% increase in the size of target lesions with an absolute increase of at least 5 mm, unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions.
  Per protocol, participants in Phase 1b receiving the Phase 2 RP2D and participants in Phase 2 RP2D were analyzed together.
Time Frame: as for outcome 6
Population: Confirmed responders in Efficacy Evaluable Population (Phase 1b/2 RP2D): participants who received ≥ 1 dose of ibrutinib (at RP2D) in combination with ≥ 1 dose of the relevant companion drug or ibrutinib (at RP2D) for the single-agent therapy and: 1) Had measurable disease per RECIST 1.1 guidelines at baseline. 2) Had ≥ 1 adequate post-baseline overall disease assessment per RECIST 1.1 guidelines.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab | Cohort 5 (UC): Ibrutinib 840 mg | Cohort 6 (UC): Ibrutinib 560 mg + Pembrolizumab
Number analyzed (Participants) | 1 | 15 | 7 | 7 | 2 | 5
months | 3.1 [NA to NA] — 1 participant analyzed | 4.4 [3.1 to 6.8] | 5.5 [3.0 to 18.0] | 11.1 [4.2 to 12.5] | 3.5 [3.1 to NA] — Not estimable because of the small number of events. | NA [2.6 to NA] — Not estimable because of the small number of events.

11. Secondary Outcome: Phase 1b: Observed Maximum Concentration (Cmax) for Ibrutinib and Its Metabolite PCI-45227 in Cohorts 1 to 4
Description: Actual collection times relative to ibrutinib administration were used for the calculation of pharmacokinetic parameters of ibrutinib and PCI-45227. For actual predose collection times that were < 0, these values were set equal to 0. Predose concentrations were applied as 24 hour concentrations in order to calculate steady-state (Cycle 2 Day 1) pharmacokinetic parameters for ibrutinib and PCI-45227. The Cmax was noted as observed.
Time Frame: Cycle 2 Day 1: predose, 1 h ± 15 min, 2 h ± 15 min, 4 h ± 15 min, 6 h ± 15 min postdose
Population: Participants with an evaluable pharmacokinetic (PK) sample for this analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 (RCC): Ibrutinib 560 mg + Everolimus | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 560 mg + Paclitaxel | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 560 mg + Cetuximab | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab
Number analyzed (Participants) | 6 | 24 | 10 | 35 | 30 | 6 | 37
ng/mL
  Ibrutininb | 172 (188) | 351 (247) | 260 (287) | 424 (319) | 164 (193) | 172 (116) | 371 (270)
  PCI-45227 | 51.2 (50.0) | 147 (77.6) | 127 (74.0) | 198 (106) | 106 (64.6) | 154 (76.1) | 177 (98.9)

12. Secondary Outcome: Phase 1b: Time to Cmax (Tmax) for Ibrutinib and Its Metabolite PCI-45227 in Cohorts 1 to 4
Description: Actual collection times relative to ibrutinib administration were used for the calculation of pharmacokinetic parameters of ibrutinib and PCI-45227. For actual predose collection times that were < 0, these values were set equal to 0. Predose concentrations were applied as 24 hour concentrations in order to calculate steady-state (Cycle 2 Day 1) pharmacokinetic parameters for ibrutinib and PCI-45227. The tmax was noted as observed.
Time Frame: Cycle 2 Day 1: predose, 1 h ± 15 min, 2 h ± 15 min, 4 h ± 15 min, 6 h ± 15 min postdose
Population: Participants with an evaluable PK sample for this analysis
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 (RCC): Ibrutinib 560 mg + Everolimus | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 560 mg + Paclitaxel | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 560 mg + Cetuximab | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab
Number analyzed (Participants) | 6 | 24 | 10 | 35 | 30 | 6 | 37
hours
  Ibrutininb | 3.01 [1.03 to 4.00] | 2.00 [0.933 to 5.90] | 3.71 [1.00 to 6.00] | 4.00 [0.833 to 6.00] | 3.89 [0.917 to 6.10] | 2.89 [1.00 to 4.08] | 2.03 [0.967 to 24.0]
  PCI-45227 | 3.03 [1.03 to 6.02] | 3.93 [1.00 to 5.90] | 4.00 [2.00 to 6.00] | 4.00 [1.00 to 6.00] | 4.00 [0.917 to 6.10] | 2.99 [1.25 to 4.08] | 4.00 [0.967 to 24.0]

13. Secondary Outcome: Phase 1b: Time of Last Observed Concentration (Tlast) for Ibrutinib and Its Metabolite PCI-45227 in Cohorts 1 to 4
Description: Actual collection times relative to ibrutinib administration were used for the calculation of pharmacokinetic parameters of ibrutinib and PCI-45227. For actual predose collection times that were < 0, these values were set equal to 0. Predose concentrations were applied as 24 hour concentrations in order to calculate steady-state (Cycle 2 Day 1) pharmacokinetic parameters for ibrutinib and PCI-45227. The tlast was noted as observed.
Time Frame: Cycle 2 Day 1: predose, 1 h ± 15 min, 2 h ± 15 min, 4 h ± 15 min, 6 h ± 15 min postdose
Population: Participants with an evaluable PK sample for this analysis
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 (RCC): Ibrutinib 560 mg + Everolimus | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 560 mg + Paclitaxel | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 560 mg + Cetuximab | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab
Number analyzed (Participants) | 6 | 24 | 10 | 34 | 29 | 5 | 37
hours
  Ibrutininb | 15.0 [5.92 to 24.0] | 24.0 [24.0 to 24.0] | 24.0 [6.00 to 24.0] | 24.0 [5.50 to 24.0] | 24.0 [5.75 to 24.0] | 24.0 [5.80 to 24.0] | 24.0 [5.42 to 24.0]
  PCI-45227 | 15.0 [5.92 to 24.0] | 24.0 [24.0 to 24.0] | 24.0 [6.00 to 24.0] | 24.0 [5.50 to 24.0] | 24.0 [5.85 to 24.0] | 24.0 [24.0 to 24.0] | 24.0 [5.75 to 24.0]

14. Secondary Outcome: Phase 1b: Area Under the Concentration-Time Curve From Time 0 to Hour 24 (AUC0-24h) for Ibrutinib and Its Metabolite PCI-45227 in Cohorts 1 to 4
Description: Actual collection times relative to ibrutinib administration were used for the calculation of pharmacokinetic parameters of ibrutinib and PCI-45227. For actual predose collection times that were < 0, these values were set equal to 0. Predose concentrations were applied as 24 hour concentrations in order to calculate steady-state (Cycle 2 Day 1) pharmacokinetic parameters for ibrutinib and PCI-45227. The AUC0-24h was calculated by the linear trapezoidal method.
Time Frame: Cycle 2 Day 1: predose, 1 h ± 15 min, 2 h ± 15 min, 4 h ± 15 min, 6 h ± 15 min postdose
Population: Participants with an evaluable PK sample for this analysis
Measure: Mean (Standard Deviation); unit: ng∙h/mL
Arm/Group | Cohort 1 (RCC): Ibrutinib 560 mg + Everolimus | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 560 mg + Paclitaxel | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 560 mg + Cetuximab | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab
Number analyzed (Participants) | 6 | 24 | 10 | 34 | 29 | 5 | 37
ng∙h/mL
  Ibrutininb | 1467 (1793) | 2568 (1968) | 2194 (3023) | 3503 (2613) | 1253 (1232) | 980 (371) | 2807 (1955)
  PCI-45227 | 646 (698) | 1810 (945) | 1146 (786) | 2604 (1435) | 1254 (777) | 1527 (717) | 2178 (1278)

15. Secondary Outcome: Phase 1b: Area Under the Concentration-Time Curve to Last Observed Time Point (AUClast) for Ibrutinib and Its Metabolite PCI-45227 in Cohorts 1 to 4
Description: Actual collection times relative to ibrutinib administration were used for the calculation of pharmacokinetic parameters of ibrutinib and PCI-45227. For actual predose collection times that were < 0, these values were set equal to 0. Predose concentrations were applied as 24 hour concentrations in order to calculate steady-state (Cycle 2 Day 1) pharmacokinetic parameters for ibrutinib and PCI-45227. The AUClast was calculated by the linear trapezoidal method.
Time Frame: Cycle 2 Day 1: predose, 1 h ± 15 min, 2 h ± 15 min, 4 h ± 15 min, 6 h ± 15 min postdose
Population: Participants with an evaluable PK sample for this analysis
Measure: Mean (Standard Deviation); unit: ng∙h/mL
Arm/Group | Cohort 1 (RCC): Ibrutinib 560 mg + Everolimus | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 560 mg + Paclitaxel | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 560 mg + Cetuximab | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab
Number analyzed (Participants) | 6 | 24 | 10 | 34 | 29 | 5 | 37
ng∙h/mL
  Ibrutininb | 1316 (1850) | 2568 (1968) | 1180 (925) | 3227 (2452) | 1107 (1178) | 847 (310) | 2647 (1967)
  PCI-45227 | 548 (741) | 1810 (945) | 859 (744) | 2380 (1561) | 1165 (803) | 1527 (717) | 2178 (1278)

16. Secondary Outcome: Phase 1b: Terminal Elimination Half-Life (t1/2term) for Ibrutinib and Its Metabolite PCI-45227 in Cohorts 1 to 4
Description: Actual collection times relative to ibrutinib administration were used for the calculation of pharmacokinetic parameters of ibrutinib and PCI-45227. For actual predose collection times that were < 0, these values were set equal to 0. Predose concentrations were applied as 24 hour concentrations in order to calculate steady-state (Cycle 2 Day 1) pharmacokinetic parameters for ibrutinib and PCI-45227. The apparent t1/2term was calculated by ln(2)/λz, where λz is the apparent elimination rate constant obtained by linear regression of three or more log-transformed data points in the terminal phase (not including Cmax).
Time Frame: Cycle 2 Day 1: predose, 1 h ± 15 min, 2 h ± 15 min, 4 h ± 15 min, 6 h ± 15 min postdose
Population: Participants with an evaluable PK sample for this analysis
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 (RCC): Ibrutinib 560 mg + Everolimus | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 560 mg + Paclitaxel | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 560 mg + Cetuximab | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab
Number analyzed (Participants) | 1 | 10 | 2 | 7 | 10 | 2 | 14
hours
  Ibrutininb: number analyzed (Participants) | 1 | 10 | 2 | 7 | 10 | 1 | 14
  Ibrutininb | NA (NA) — Not determined due to insufficient data. | 6.28 (2.35) | 7.24 (2.36) | 4.31 (1.95) | 5.54 (1.75) | NA (NA) — Not determined due to insufficient data. | 5.52 (1.26)
  PCI-45227: number analyzed (Participants) | 1 | 4 | 2 | 4 | 9 | 2 | 14
  PCI-45227 | NA (NA) — Not determined due to insufficient data. | 8.00 (0.489) | 5.08 (0.304) | 6.79 (4.38) | 6.48 (2.11) | 8.10 (NA) — Not determined due to insufficient data. | 8.02 (2.17)

17. Secondary Outcome: Phase 1b: Terminal Elimination Rate Constant (λz) for Ibrutinib and Its Metabolite PCI-45227 in Cohorts 1 to 4
Description: Actual collection times relative to ibrutinib administration were used for the calculation of pharmacokinetic parameters of ibrutinib and PCI-45227. For actual predose collection times that were < 0, these values were set equal to 0. Predose concentrations were applied as 24 hour concentrations in order to calculate steady-state (Cycle 2 Day 1) pharmacokinetic parameters for ibrutinib and PCI-45227. The λz is the apparent elimination rate constant obtained by linear regression of three or more log-transformed data points in the terminal phase (not including Cmax).
Time Frame: Cycle 2 Day 1: predose, 1 h ± 15 min, 2 h ± 15 min, 4 h ± 15 min, 6 h ± 15 min postdose
Population: Participants with an evaluable PK sample for this analysis
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Cohort 1 (RCC): Ibrutinib 560 mg + Everolimus | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 560 mg + Paclitaxel | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 560 mg + Cetuximab | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab
Number analyzed (Participants) | 1 | 10 | 2 | 7 | 10 | 2 | 14
1/h
  Ibrutininb: number analyzed (Participants) | 1 | 10 | 2 | 7 | 10 | 1 | 14
  Ibrutininb | NA (NA) — Not determined due to insufficient data. | 0.125 (0.0477) | 0.101 (0.0327) | 0.195 (0.0902) | 0.135 (0.0349) | NA (NA) — Not determined due to insufficient data. | 0.132 (0.0296)
  PCI-45227: number analyzed (Participants) | 0 | 4 | 2 | 4 | 9 | 2 | 8
  PCI-45227 |  | 0.0870 (0.00535) | 0.137 (0.00849) | 0.149 (0.103) | 0.118 (0.0399) | 0.0897 (NA) — Not determined due to insufficient data. | 0.0942 (0.0336)

18. Secondary Outcome: Phase 1b: Apparent Total Clearance at Steady-State (CLss/F) for Ibrutinib in Cohorts 1 to 4
Description: Actual collection times relative to ibrutinib administration were used for the calculation of pharmacokinetic parameters of ibrutinib and PCI-45227. For actual predose collection times that were < 0, these values were set equal to 0. Predose concentrations were applied as 24 hour concentrations in order to calculate steady-state (Cycle 2 Day 1) pharmacokinetic parameters for ibrutinib and PCI-45227. Apparent total CLss/F (Cycle 2 Day 1) was calculated as dose/AUC0-24h.
Time Frame: Cycle 2 Day 1: predose, 1 h ± 15 min, 2 h ± 15 min, 4 h ± 15 min, 6 h ± 15 min postdose
Population: Participants with an evaluable PK sample for this analysis
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort 1 (RCC): Ibrutinib 560 mg + Everolimus | Cohort 1 (RCC): Ibrutinib 840 mg + Everolimus | Cohort 2 (UC): Ibrutinib 560 mg + Paclitaxel | Cohort 2 (UC): Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CRC): Ibrutinib 560 mg + Cetuximab | Cohort 4 (CRC): Ibrutinib 840 mg + Cetuximab
Number analyzed (Participants) | 6 | 24 | 10 | 34 | 29 | 5 | 37
L/h | 1103 (1370) | 622 (647) | 994 (1217) | 1067 (2742) | 1102 (1412) | 645 (248) | 595 (726)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Maximum time on study (Phase 1b/2 RP2D) was 37.4 months, 44.7 months, 41.9 months, 23.5 months, 17.3 months, 20.1 months for Cohorts 1, 2, 3, 4, 5, 6 respectively. Serious/Other Adverse Events: First dose of study drug to end of treatment + 30 days. Mean time on treatment was: 14.5, 20.1, 16.3, 13.5, 12.8, 11.0, 10.9, 10.4, 15.8, 8.8, 13.5, 7.7, 8.4, 7.8, 9.2 months for the Reporting Groups presented below (from left to right), respectively.
Description: A participant is 'at risk' in Phase 1b if they were enrolled in Phase 1b. A participant is 'at risk' in Phase 2 if they were enrolled in Phase 2 or if they were enrolled in Phase 1b and discontinued the study after the start of Phase 2 date (defined as the date for first Phase 2 participant was enrolled for that cohort). Therefore, a participant adverse event could be double counted if the participant was in Phase 1b and then continued to Phase 2 dosing at that cohort.
Groups:
- Cohort 1 (RCC) Phase 1b: Ibrutinib 560 mg + Everolimus: Participants with RCC in Phase 1b received ibrutinib 560 mg QD in combination with everolimus 10 mg QD.
- Cohort 1 (RCC) Phase 1b: Ibrutinib 840 mg + Everolimus: Participants with RCC in Phase 1b received ibrutinib 840 mg QD in combination with everolimus 10 mg QD.
- Cohort 1 (RCC) Phase 2: Ibrutinib 840 mg + Everolimus: Participants with RCC in Phase 2 received ibrutinib 840 mg QD in combination with everolimus 10 mg QD.
- Cohort 2 (UC) Phase 1b: Ibrutinib 560 mg + Paclitaxel: Participants with UC in Phase 1b received ibrutinib 560 mg QD in combination with paclitaxel 80 mg/m^2, once weekly, in continual 3 weekly cycles.
- Cohort 2 (UC) Phase 1b: Ibrutinib 840 mg + Paclitaxel: Participants with UC in Phase 1b received ibrutinib 840 mg QD in combination with paclitaxel 80 mg/m^2, once weekly, in continual 3 weekly cycles.
- Cohort 2 (UC) Phase 2: Ibrutinib 840 mg + Paclitaxel: Participants with UC in Phase 2 received ibrutinib 840 mg QD in combination with paclitaxel 80 mg/m^2, once weekly, in continual 3 weekly cycles.
- Cohort 3 (GA) Phase 1b: Ibrutinib 560 mg + Docetaxel: Participants with GA in Phase 1b received ibrutinib 560 mg QD in combination with docetaxel administered as a 60 minute infusion (±10 minutes) at a dose level of 60 - 75 mg/m^2, given continually in 21 day cycles.
- Cohort 3 (GA) Phase 2 (RP2D): Ibrutinib 560 mg + Docetaxel: Participants with GA in Phase 2 received ibrutinib 560 mg QD in combination with docetaxel administered as a 60 minute infusion (±10 minutes) at a dose level of 60 - 75 mg/m^2, given continually in 21 day cycles.
- Cohort 4 (CA) Phase 1b: Ibrutinib 560 mg + Cetuximab: Participants with CRC in Phase 1b received ibrutinib 560 mg QD in combination with cetuximab 400 mg/m^2 administered as a 120-minute IV infusion. Subsequent weekly dose (all other infusions) was 250 mg/m^2 infused over 60 minutes.
- Cohort 4 (CA) Phase 1b: Ibrutinib 840 mg + Cetuximab: Participants with CRC in Phase 1b received ibrutinib 840 mg QD in combination with cetuximab 400 mg/m^2 administered as a 120-minute IV infusion. Subsequent weekly dose (all other infusions) was 250 mg/m^2 infused over 60 minutes.
- Cohort 4 (CA) Phase 2 (RP2D): Ibrutinib 840 mg + Cetuximab: Participants with CRC in Phase 2 received ibrutinib 840 mg QD in combination with cetuximab 400 mg/m^2 administered as a 120-minute IV infusion. Subsequent weekly dose (all other infusions) was 250 mg/m^2 infused over 60 minutes.
- Cohort 5 (UC) Phase 1b: Ibrutinib 840 mg: Participants with UC in Phase 1b received monotherapy with ibrutinib 840 mg QD.
- Cohort 5 (UC) Phase 2: Ibrutinib 840 mg: Participants with UC in Phase 2 received monotherapy with ibrutinib 840 mg QD.
- Cohort 6 (UC) Phase 1b: Ibrutinib 560 mg + Pembrolizumab: Participants with UC in Phase 1b received ibrutinib 560 mg QD in combination with pembrolizumab 200 mg IV every 3 weeks.
- Cohort 6 (UC) Phase 2: Ibrutinib 560 mg + Pembrolizumab: Participants with UC in Phase 2 received ibrutinib 560 mg QD in combination with pembrolizumab 200 mg IV every 3 weeks.
Arm/Group | Cohort 1 (RCC) Phase 1b: Ibrutinib 560 mg + Everolimus | Cohort 1 (RCC) Phase 1b: Ibrutinib 840 mg + Everolimus | Cohort 1 (RCC) Phase 2: Ibrutinib 840 mg + Everolimus | Cohort 2 (UC) Phase 1b: Ibrutinib 560 mg + Paclitaxel | Cohort 2 (UC) Phase 1b: Ibrutinib 840 mg + Paclitaxel | Cohort 2 (UC) Phase 2: Ibrutinib 840 mg + Paclitaxel | Cohort 3 (GA) Phase 1b: Ibrutinib 560 mg + Docetaxel | Cohort 3 (GA) Phase 2 (RP2D): Ibrutinib 560 mg + Docetaxel | Cohort 4 (CA) Phase 1b: Ibrutinib 560 mg + Cetuximab | Cohort 4 (CA) Phase 1b: Ibrutinib 840 mg + Cetuximab | Cohort 4 (CA) Phase 2 (RP2D): Ibrutinib 840 mg + Cetuximab | Cohort 5 (UC) Phase 1b: Ibrutinib 840 mg | Cohort 5 (UC) Phase 2: Ibrutinib 840 mg | Cohort 6 (UC) Phase 1b: Ibrutinib 560 mg + Pembrolizumab | Cohort 6 (UC) Phase 2: Ibrutinib 560 mg + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 3/3 | 1/7 | 22/38 | 3/4 | 4/10 | 51/55 | 13/21 | 17/31 | 6/8 | 4/12 | 31/44 | 2/10 | 20/33 | 4/17 | 3/13
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/7 | 18/38 | 2/4 | 5/10 | 32/55 | 15/21 | 12/31 | 5/8 | 2/12 | 14/44 | 3/10 | 16/33 | 7/17 | 3/13
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 34/38 | 4/4 | 10/10 | 51/55 | 20/21 | 26/31 | 8/8 | 12/12 | 40/44 | 9/10 | 29/33 | 16/17 | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (RCC) Phase 1b: Ibrutinib 560 mg + Everolimus (N=3) | Cohort 1 (RCC) Phase 1b: Ibrutinib 840 mg + Everolimus (N=7) | Cohort 1 (RCC) Phase 2: Ibrutinib 840 mg + Everolimus (N=38) | Cohort 2 (UC) Phase 1b: Ibrutinib 560 mg + Paclitaxel (N=4) | Cohort 2 (UC) Phase 1b: Ibrutinib 840 mg + Paclitaxel (N=10) | Cohort 2 (UC) Phase 2: Ibrutinib 840 mg + Paclitaxel (N=55) | Cohort 3 (GA) Phase 1b: Ibrutinib 560 mg + Docetaxel (N=21) | Cohort 3 (GA) Phase 2 (RP2D): Ibrutinib 560 mg + Docetaxel (N=31) | Cohort 4 (CA) Phase 1b: Ibrutinib 560 mg + Cetuximab (N=8) | Cohort 4 (CA) Phase 1b: Ibrutinib 840 mg + Cetuximab (N=12) | Cohort 4 (CA) Phase 2 (RP2D): Ibrutinib 840 mg + Cetuximab (N=44) | Cohort 5 (UC) Phase 1b: Ibrutinib 840 mg (N=10) | Cohort 5 (UC) Phase 2: Ibrutinib 840 mg (N=33) | Cohort 6 (UC) Phase 1b: Ibrutinib 560 mg + Pembrolizumab (N=17) | Cohort 6 (UC) Phase 2: Ibrutinib 560 mg + Pembrolizumab (N=13)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 7 (10) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERICARDITIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PLEUROPERICARDITIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ILEUS PARALYTIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MELAENA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENERALISED OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUDDEN CARDIAC DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUDDEN DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AMYLOIDOSIS (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATYPICAL PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BILIARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EMPHYSEMATOUS CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES SIMPLEX (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
KLEBSIELLA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENINGITIS ASEPTIC (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARONYCHIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (3) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SOFT TISSUE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URETERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 6 (12) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UROSEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT STOMA COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD URINE PRESENT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOPHAGIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NECK MASS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLORECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
METASTASES TO SPINE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RADICULOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
BLADDER PAIN (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RENAL INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URETHRAL STENOSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY ARTERY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLEURODESIS (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (RCC) Phase 1b: Ibrutinib 560 mg + Everolimus (N=3) | Cohort 1 (RCC) Phase 1b: Ibrutinib 840 mg + Everolimus (N=7) | Cohort 1 (RCC) Phase 2: Ibrutinib 840 mg + Everolimus (N=38) | Cohort 2 (UC) Phase 1b: Ibrutinib 560 mg + Paclitaxel (N=4) | Cohort 2 (UC) Phase 1b: Ibrutinib 840 mg + Paclitaxel (N=10) | Cohort 2 (UC) Phase 2: Ibrutinib 840 mg + Paclitaxel (N=55) | Cohort 3 (GA) Phase 1b: Ibrutinib 560 mg + Docetaxel (N=21) | Cohort 3 (GA) Phase 2 (RP2D): Ibrutinib 560 mg + Docetaxel (N=31) | Cohort 4 (CA) Phase 1b: Ibrutinib 560 mg + Cetuximab (N=8) | Cohort 4 (CA) Phase 1b: Ibrutinib 840 mg + Cetuximab (N=12) | Cohort 4 (CA) Phase 2 (RP2D): Ibrutinib 840 mg + Cetuximab (N=44) | Cohort 5 (UC) Phase 1b: Ibrutinib 840 mg (N=10) | Cohort 5 (UC) Phase 2: Ibrutinib 840 mg (N=33) | Cohort 6 (UC) Phase 1b: Ibrutinib 560 mg + Pembrolizumab (N=17) | Cohort 6 (UC) Phase 2: Ibrutinib 560 mg + Pembrolizumab (N=13)
ANAEMIA (Blood and lymphatic system disorders) | 2 (5) | 2 (16) | 19 (58) | 1 (1) | 4 (7) | 20 (57) | 8 (32) | 16 (33) | 1 (1) | 1 (1) | 5 (9) | 0 (0) | 6 (12) | 0 (0) | 0 (0)
COAGULOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INCREASED TENDENCY TO BRUISE (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 3 (14) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 8 (11) | 9 (15) | 7 (27) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPONTANEOUS HAEMATOMA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 3 (5) | 8 (23) | 0 (0) | 2 (5) | 3 (5) | 4 (10) | 4 (6) | 1 (2) | 1 (1) | 6 (10) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DRY EYE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE DISORDER (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LACRIMATION INCREASED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISUAL ACUITY REDUCED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VITREOUS DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 6 (6) | 2 (5) | 5 (7) | 0 (0) | 1 (1) | 5 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 6 (10) | 0 (0) | 2 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHANGE OF BOWEL HABIT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 5 (6) | 14 (15) | 5 (7) | 5 (6) | 1 (1) | 2 (2) | 7 (7) | 1 (1) | 8 (11) | 7 (7) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (3) | 5 (17) | 16 (30) | 4 (14) | 8 (17) | 36 (89) | 14 (34) | 10 (20) | 2 (3) | 6 (8) | 19 (35) | 0 (0) | 10 (14) | 8 (8) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 2 (14) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 6 (6) | 3 (5) | 2 (2) | 0 (0) | 0 (0) | 8 (9) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL TRACT IRRITATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
GLOSSODYNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIP OEDEMA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIP PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
MELAENA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 13 (32) | 0 (0) | 6 (9) | 17 (28) | 12 (20) | 5 (8) | 4 (4) | 2 (4) | 12 (15) | 5 (5) | 12 (14) | 5 (6) | 1 (1)
OESOPHAGEAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL MUCOSAL ERYTHEMA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAROTID GLAND ENLARGEMENT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 2 (3) | 3 (6) | 20 (50) | 1 (1) | 3 (6) | 14 (22) | 9 (17) | 8 (9) | 4 (4) | 5 (6) | 20 (44) | 0 (0) | 3 (3) | 4 (8) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 2 (4) | 8 (14) | 1 (5) | 3 (4) | 14 (21) | 10 (18) | 5 (6) | 2 (2) | 1 (1) | 8 (12) | 4 (5) | 6 (10) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 1 (2) | 3 (13) | 8 (17) | 1 (1) | 3 (13) | 27 (112) | 2 (3) | 9 (36) | 1 (2) | 4 (4) | 5 (13) | 1 (2) | 11 (17) | 0 (0) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHILLS (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 3 (4) | 14 (27) | 3 (5) | 5 (13) | 15 (30) | 8 (37) | 8 (12) | 2 (2) | 8 (13) | 14 (27) | 1 (1) | 9 (13) | 6 (10) | 4 (5)
GAIT DISTURBANCE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
LOCALISED OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NODULE (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 2 (5) | 0 (0) | 8 (8) | 2 (2) | 1 (1) | 14 (20) | 4 (5) | 2 (2) | 4 (5) | 3 (4) | 4 (6) | 2 (2) | 4 (4) | 3 (5) | 0 (0)
PAIN (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 2 (6) | 6 (6) | 0 (0) | 1 (2) | 15 (24) | 4 (5) | 4 (5) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 2 (4) | 3 (3) | 0 (0)
SWELLING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SWELLING FACE (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THIRST (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 5 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOLLICULITIS (Infections and infestations) | 0 (0) | 1 (1) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FUNGAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FURUNCLE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIP INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PARONYCHIA (Infections and infestations) | 0 (0) | 1 (2) | 5 (8) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 1 (1) | 2 (2) | 4 (11) | 14 (24) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROSTATITIS ESCHERICHIA COLI (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PSEUDOMONAS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 5 (9) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 4 (5) | 1 (1) | 4 (4) | 1 (1) | 2 (3)
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WOUND HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (7) | 1 (2) | 3 (13) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (4) | 1 (1) | 3 (9) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 0 (0)
BLOOD BICARBONATE DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 2 (14) | 1 (2) | 7 (20) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
BLOOD IRON DECREASED (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD MAGNESIUM DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD POTASSIUM DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
BLOOD UREA INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
BLOOD URINE PRESENT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (7) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 1 (2) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 9 (11) | 2 (5) | 8 (18) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 1 (2) | 5 (7) | 0 (0) | 1 (1) | 6 (10) | 2 (2) | 4 (6) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
PROTEIN URINE PRESENT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RED BLOOD CELLS URINE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 1 (2) | 4 (5) | 0 (0) | 2 (2) | 0 (0) | 7 (8) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (12) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 4 (9) | 13 (21) | 2 (4) | 7 (17) | 18 (33) | 8 (19) | 10 (19) | 3 (3) | 5 (8) | 9 (13) | 4 (5) | 8 (10) | 1 (1) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (7) | 5 (14) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 6 (8) | 7 (9) | 2 (2) | 3 (4) | 1 (1) | 6 (16) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 1 (1) | 5 (9) | 3 (5) | 1 (2) | 3 (5) | 1 (1) | 9 (22) | 0 (0) | 3 (4) | 2 (2) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (8) | 1 (1) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3) | 6 (7) | 2 (3) | 1 (2) | 11 (18) | 6 (6) | 3 (8) | 1 (2) | 2 (3) | 2 (4) | 0 (0) | 2 (3) | 6 (7) | 2 (5)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 10 (12) | 1 (2) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ENTHESOPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (5) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (4) | 5 (5) | 4 (7) | 2 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 1 (2) | 4 (4) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 2 (2) | 0 (0) | 2 (3)
CEREBRAL DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 9 (11) | 1 (1) | 0 (0) | 10 (15) | 5 (8) | 2 (2) | 0 (0) | 1 (1) | 5 (6) | 1 (1) | 8 (12) | 4 (4) | 0 (0)
DYSAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 6 (10) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
HEAD DISCOMFORT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (2) | 3 (5) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MYOCLONUS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEUROTOXICITY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (31) | 0 (0) | 7 (19) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL SENSORIMOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (2) | 14 (29) | 6 (11) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TASTE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (15) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
DISORIENTATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (4) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 5 (7) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
PANIC ATTACK (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 10 (14) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 4 (7) | 1 (1)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 1 (9) | 4 (5) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 (0) | 1 (11) | 3 (6) | 0 (0) | 0 (0) | 4 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
BALANOPOSTHITIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERINEAL ERYTHEMA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 11 (14) | 0 (0) | 1 (1) | 4 (4) | 5 (13) | 1 (1) | 1 (2) | 2 (2) | 5 (5) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (7) | 4 (4) | 0 (0) | 1 (2) | 8 (11) | 3 (5) | 0 (0) | 2 (4) | 1 (1) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 21 (31) | 1 (2) | 2 (2) | 7 (9) | 1 (1) | 4 (6) | 0 (0) | 2 (2) | 9 (12) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OROPHARYNGEAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PAINFUL RESPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPUTUM DISCOLOURED (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 3 (3) | 15 (21) | 6 (9) | 8 (8) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 5 (8) | 1 (1) | 1 (1) | 6 (8) | 1 (1) | 2 (2) | 4 (16) | 8 (16) | 31 (130) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (3) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 20 (37) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAIR COLOUR CHANGES (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIRSUTISM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAIL TOXICITY (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ONYCHALGIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ONYCHOMADESIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 12 (30) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 7 (14) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
PIGMENTATION DISORDER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (9) | 0 (0) | 0 (0) | 4 (5) | 6 (6) | 2 (2) | 2 (4) | 3 (4) | 14 (21) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
PURPURA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (4) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 3 (6) | 0 (0) | 2 (4) | 1 (1) | 0 (0)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 9 (31) | 0 (0) | 0 (0) | 5 (10) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 7 (24) | 0 (0) | 2 (2) | 4 (8) | 2 (4)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 2 (13) | 2 (7) | 0 (0) | 1 (1) | 3 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
JUGULAR VEIN DISTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PALLOR (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT02599324/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/24/NCT02599324/SAP_001.pdf